CLINICAL TRIAL: NCT04264065
Title: Albumin and Prognosis of Severely Burned Patients Retrospective, Prospective, Observational Study for the BurnICU Group of ESICM
Brief Title: Albumin and Prognosis of Severely Patients Burns
Acronym: ALBUBURN
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: TPS1122427
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Severe Burn
Keywords: Severe Burn; acute respiratory distress; acute kidney injury; Albumin
MeSH Terms: conditions — Burns; Acute Lung Injury; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hemodynamic management has long been identified as a key factor affecting burn prognosis. However, large amounts of crystalloid infusion have been associated with the development or aggravation of organ failure (acute respiratory distress syndrome, vascular injury, acute renal failure, and intra-abdominal hypertension) which worsens the final prognosis.

The use of albumin during the first 24 hours of burn resuscitation is controversial since capillary leakage may cause transcapillary passage of large molecules into the interstitial space. In fact, human albumin has multiple physiological effects, including regulation of colloidal osmotic pressure, antioxidant properties, nitric oxide modulation and buffering capacities, plasma binding and transport of various substances, which may be particularly important in severe burns.

Currently available data suggest that administration of exogenous albumin during the first 24 hours of resuscitation of severe burn patients may be associated with improved outcomes. Multi-centre randomized controlled trials with adequate power should be undertaken in burned patients.

DETAILED DESCRIPTION:
In the participating centers: severe burn adult patients with a TBSA burn >30% will be included and followed for 90 days after admission. This observational study will allow us to collect and analyze data in order to design a quality interventional trial evaluating the value of albumin in the initial management of the severely burned patient.

The primary objective of the study is to describe the incidence of a combined endpoint of mortality, severe acute renal failure (stage 3) and severe acute respiratory distress syndrome in severely burned patients.

Secondary Objectives

1. Describe the prognosis of patients with severe burns, with particular emphasis on the impact of albumin on the prognosis of patients with severe burns.
2. Describe how albumin is administered (i.e. doses, duration of treatment, continuous vs. bolus administration, hyperoncotic vs. hypooncotic solutions, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Burns > 30% SCT
* Patients admitted to the ICU within 12 hours of a burn.

Exclusion Criteria:

* Pregnancy
* Patients with a limitation of active therapeutics on admission to BICU
* Pre-hospital cardiac arrest
* Moribund patients: pre-hospital cardiac arrest, CBS burn >95%.
* Age >80 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: it is a population of adults burned to more than 30% of total skin surface. In fact, beyond this surface, the investigators expect to observe a large volume of perfused crystalloid and potentially an incidence of the primary endpoint of around 40%. These are the people who could potentially benefit the most from albumin therapy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-09-16 (Actual); Primary Completion 2027-01-16 (Estimated); Study Completion 2027-01-16 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be a combined endpoint of mortality, stage 3 acute renal failure and severe acute respiratory distress syndrome within 28 days of burn injury. | 28 days of burn injury

SECONDARY OUTCOMES:
Rate of patients with acute renal failure on days 28 and 90 | days 28 and 90 of burn injury
  Kidney disease improving global outcome (KDIGO) definition
Rate of patients with Acute respiratory distress syndrome (ARDS) on days 28 and 90 | days 28 and 90 of burn injury
  Berlin Definition
Rate of patients with Acute Abdominal Compartment Syndrome | days 28 and 90 of burn injury
  ACS is defined as sustained AIP > 20 mmHg associated with new or ongoing organ dysfunction or failure
Rate of patients with Sepsis and septic shock | Days 28 and 90
  Definition of Sepsis 3
SOFA Score | between Day 1 and Day 7
  Sepsis related organ failure assessment (SOFA) score the minimum value is 0 meaning no organ dysfunction and the maximum being 24 meaning the maximum organs dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: François Dr DEPRET, MD, Principal Investigator — Hospital Saint Louis (AP-HP)
Locations (1):
- Hopital saint Louis, Paris, France, France

REFERENCES:
- [Background] Arlati S, Storti E, Pradella V, Bucci L, Vitolo A, Pulici M. Decreased fluid volume to reduce organ damage: a new approach to burn shock resuscitation? A preliminary study. Resuscitation. 2007 Mar;72(3):371-8. doi: 10.1016/j.resuscitation.2006.07.010. Epub 2006 Nov 29. PMID 17137702
- [Background] Mason SA, Nathens AB, Finnerty CC, Gamelli RL, Gibran NS, Arnoldo BD, Tompkins RG, Herndon DN, Jeschke MG; Inflammation and the Host Response to Injury Collaborative Research Program.. Hold the Pendulum: Rates of Acute Kidney Injury are Increased in Patients Who Receive Resuscitation Volumes Less than Predicted by the Parkland Equation. Ann Surg. 2016 Dec;264(6):1142-1147. doi: 10.1097/SLA.0000000000001615. PMID 27828823
- [Background] Soussi S, Taccori M, De Tymowski C, Depret F, Chaussard M, Fratani A, Jully M, Cupaciu A, Ferry A, Benyamina M, Serror K, Boccara D, Chaouat M, Mimoun M, Cattan P, Zagdanski AM, Anstey J, Mebazaa A, Legrand M; PRONOBURN group. Risk Factors for Acute Mesenteric Ischemia in Critically Ill Burns Patients-A Matched Case-Control Study. Shock. 2019 Feb;51(2):153-160. doi: 10.1097/SHK.0000000000001140. PMID 29561390
- [Background] Klein MB, Hayden D, Elson C, Nathens AB, Gamelli RL, Gibran NS, Herndon DN, Arnoldo B, Silver G, Schoenfeld D, Tompkins RG. The association between fluid administration and outcome following major burn: a multicenter study. Ann Surg. 2007 Apr;245(4):622-8. doi: 10.1097/01.sla.0000252572.50684.49. PMID 17414612
- [Background] Markell KW, Renz EM, White CE, Albrecht ME, Blackbourne LH, Park MS, Barillo DA, Chung KK, Kozar RA, Minei JP, Cohn SM, Herndon DN, Cancio LC, Holcomb JB, Wolf SE. Abdominal complications after severe burns. J Am Coll Surg. 2009 May;208(5):940-7; discussion 947-9. doi: 10.1016/j.jamcollsurg.2008.12.023. Epub 2009 Mar 26. PMID 19476867
- [Background] Cooper AB, Cohn SM, Zhang HS, Hanna K, Stewart TE, Slutsky AS; ALBUR Investigators. Five percent albumin for adult burn shock resuscitation: lack of effect on daily multiple organ dysfunction score. Transfusion. 2006 Jan;46(1):80-9. doi: 10.1111/j.1537-2995.2005.00667.x. PMID 16398734
- [Background] Cochran A, Morris SE, Edelman LS, Saffle JR. Burn patient characteristics and outcomes following resuscitation with albumin. Burns. 2007 Feb;33(1):25-30. doi: 10.1016/j.burns.2006.10.005. PMID 17223485